CLINICAL TRIAL: NCT06288087
Title: Comparing Machine Guided VR Based Training With Educator Guided Training in Metaverse Environment: A Randomized Controlled Study
Brief Title: Comparing Machine Guided VR Based Training With Educator Guided Training in Metaverse
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Emin Aksoy, Associate professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-20/672
Record Dates: First submitted 2024-02-14; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Advanced Cardiac Life Support; Virtual Reality; Serious Game

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: the group trained with VR Based Training with Machine Guidance will be referred as MG group and the group trained with VR Based Training with Educators Guidance in Metaverse will be referred as EG group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MG Group (Other): The group trained with VR Based Training with Machine Guidance will be referred as MG group.
  Interventions: Other: VR Based Training with Machine Guidance (MG Group)
- EG Group (Other): The group trained with VR Based Training with Educators Guidance in Metaverse will be referred as EG group.
  Interventions: Other: VR Based Training with Educator Guidance in Metaverse (EG Group)

INTERVENTIONS:
Other: VR Based Training with Machine Guidance (MG Group) — The members of both groups will undertake a VR based basic training for ALS. Afterwards MG group were trained with VR based Advanced Training Module, which provides training with full machine guidance. The knowledge level will then be evaluated by the exam mode of the VR based training module
  Arms: MG Group
Other: VR Based Training with Educator Guidance in Metaverse (EG Group) — The members of both groupswill undertake a VR based basic training for ALS. Afterwards EG group will attend at VR based Educator guided training in metaverse. The knowledge level will then be evaluated by the exam mode of the VR based training module
  Arms: EG Group

SUMMARY:
The main aim of this study is to compare the learning outcomes of machine guided VR based training for adult advanced life support with educator guided training in metaverse environment.

DETAILED DESCRIPTION:
Online education stands as one of the metaverse's potential application areas. The metaverse's ability to offer shared social connections differs it from existing online educational platforms such as Simulation, AR, and VR, which primarily focus on presenting virtual content and environments without fostering communal interaction. This facilitates interaction between learners and educators during metaverse-based training sessions allowing educators to guide the learners and provide feedback. The educators' presence fosters communication and collaboration during training sessions, thereby enhancing learners' motivation and engagement.

In our university, a VR-based multiplayer training module within the metaverse environment specifically designed for ALS (Adult Advanced Life Support) training has been developed. This module serves as an additional training tool to simulation-based training, enabling learners to receive guidance either from machine algorithms or educators within the metaverse. The objective of this study is to reveal the benefits of educator presence in the metaverse during VR-based training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering for the study

Exclusion Criteria:

* Previously experienced VR-induced motion sickness
* Previous Advanced Life Support training
* Other medical conditions like vertigo attacks
* Being under medication, which may cause vertigo like symptoms.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-04-11 (Estimated)

PRIMARY OUTCOMES:
Comparing Learning outcome of the Advanced Cardiac Life Support Training of the two interventions used in this study | The participants will complete the exam mode for final evaluation right after the completion of training on the same day
  Knowledge assessment will be conducted using the exam mode of the VR-based training module, evaluating users' performances utilizing an international algorithm developed by the American Heart Association (AHA) and Crisis Resource Management Criteria (CRM) derived from Aviation Training Algorithms. Seventy percent of the total performance score will be derived from ACLS assessments, with the remaining percentage calculated from CRM performances of the participants. The primary outcome of the study will be determined by the total score obtained through the exam mode of the VR-based training module.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University CASE (Center of Advanced Simulation and Education), Istanbul, Non-US/Canada, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Upon request by email.
Supporting Information: Study Protocol, ICF
Time Frame: 6 Months
Access Criteria: Upon request by email.

REFERENCES:
- [Derived] Kitapcioglu D, Aksoy ME, Ozkan AE, Usseli T. Comparing Learning Outcomes of Machine-Guided Virtual Reality-Based Training With Educator-Guided Training in a Metaverse Environment: Randomized Controlled Trial. JMIR Serious Games. 2024 Aug 7;12:e58654. doi: 10.2196/58654. PMID 39110497